CLINICAL TRIAL: NCT02146209
Title: Comparative Randomized, Single Dose, Three-Period Crossover Open-Label Study to Determine the Bioequivalence Of Terix Labs Ltd Metronidazole Benzoate (400 mg Metronidazole Per Sachet Oral Granules (Formula A)) Relative to 500 mg From Sanofi-aventis Flagyl 125 mg/5 ml (125 mg Metronidazole Per 5 ml Suspension (Formula B)) and Zentiva Flagyl™ 400 mg Tablets (400 mg Metronidazole Per Film Coated Tablets (Formula C)) , After an Oral Administration to Healthy Adults Under Fasting Conditions
Brief Title: Study to Determine the Equivalence of Three Products Containing Metronidazole Benzoate.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verisfield UK Ltd. Greek Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MET-GST006
Record Dates: First submitted 2014-05-16; First posted 2014-05-23 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Benchmarking; Metronidazole; Suspensions

ARMS (3):
- Test Product Formula A (Experimental): Metronidazole benzoate
  Interventions: Drug: Metronidazole benzoate
- Reference Product Formula B (Active Comparator): Flagyl 125 mg/5 ml oral suspension
  Interventions: Drug: Flagyl 125 mg/5 ml oral suspension
- Reference Product Formula C (Active Comparator): Flagyl 400 mg Tablets
  Interventions: Drug: Flagyl 400 mg Tablets

INTERVENTIONS:
Drug: Metronidazole benzoate — Single oral dose of 400 mg
  Arms: Test Product Formula A
Drug: Flagyl 125 mg/5 ml oral suspension — Single oral dose of 500 mg (20 ml suspension)
  Arms: Reference Product Formula B
Drug: Flagyl 400 mg Tablets — Single oral dose of 400 mg
  Arms: Reference Product Formula C

SUMMARY:
The purpose of this study is to determine whether Terix Labs Ltd Metronidazole benzoate (400 mg Metronidazole Per Sachet Oral Granules) is bioequivalent to 500 mg Sanofi-aventis Flagyl 125 mg/5 ml (125 mg Metronidazole Per 5 ml Suspension) and to Zentiva Flagyl™ 400 mg Tablets (400 mg Metronidazole Per Film Coated Tablets).

DETAILED DESCRIPTION:
This study is a pilot study exploited for exploratory purposes to compare the absorption and disposition kinetics of three products containing metronidazole under fasting conditions. These products are: Metronidazole benzoate (formula A), Test product manufactured by ONE PHARMA, Greece. Flagyl 125 mg/5 ml (formula B), a Reference product manufactured by Unither Liquid Manufacturing, France and Flagyl™ 400 mg Tablets (formula C), a Reference product manufactured by Famar Health Care Services, Spain. The bioequivalence of a single 400 mg dose of products A and C, and a single 500 mg dose of product B will be assessed by comparing the pharmacokinetic parameters derived from the plasma concentration-time profiles for metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive.
* Body Mass Index (BMI) range is within 18.5 - 30 Kg/m2.
* Subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.

Exclusion Criteria:

* Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
* Results of laboratory tests are within the normal range except for Hb and RBC indices test that should be within the 5% of reference range and kidney function tests (Creatinine will be accepted if below reference range) that are outside the reference range. (Laboratory tests are performed not longer than two weeks before the initiation of the clinical study).
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject is a heavy smoker (more than 10 cigarettes per day).
* Subject does not agree not to take any prescription or non-prescription drugs within the two weeks preceding the first study drug administration until donating the last sample of the study.
* Subject does not agree not to take any vitamins taken for nutritional purposes within two days before first study drug administration until donating the last sample of the study.
* Subject is on a special diet (for example subject is a vegetarian).
* Subject consumes large quantities of alcohol or beverages containing methylxanthines e.g. caffeine (coffee, tea, cola, chocolate etc).
* Subject does not agree not to consume any beverages or food containing alcohol 48 hours prior to study drug administration until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or food containing methyl-xanthines e.g. caffeine (coffee, tea, cola, chocolate etc.) 24 hours prior to the study drug administration until the end of confinement period.
* Subject does not agree not to consume any beverages or food containing grapefruit 7 days prior to first study drug administration until donating the last sample in the study.
* Subject has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 80 days before first study drug administration.
* Subject intends to be hospitalized within 3 months after first study drugs administration.
* Subjects who donated blood or its derivatives in the past 3 months or who through completion of this study, would have donated more than 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.
* Subject has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders.
* Subject who have been engaged in strenuous exercise at least one day prior to dosing till the last sample of each respective period.
* Subject having at screening examination a pulse outside the normal range of (60-100 beat per minute) or a body temperature outside the normal range of (36.4-37.7 ○C) or a respiratory rate outside the normal range of (14-20 breath per minute) or a sitting blood pressure less than 100/60 mm Hg or more than or equal to 140/90 mm Hg.
* Subject has history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration time profiles under the curve (AUC) | 0, 15, 30 and 45 minutes and 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | 0, 15, 30 and 45 minutes and 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Maximum measured plasma concentration
Time to maximum concentration (Tmax) | 0, 15, 30 and 45 minutes and 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value
Elimination rate constant (Kel) | 0, 15, 30 and 45 minutes and 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Apparent first-order elimination or terminal rate constant
Terminal half life (t1/2) | 0, 15, 30 and 45 minutes and 1.00, 1.33, 1.67, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The elimination or terminal half-life
Number of participants with Adverse Events | 17 days
  Subjects will be monitored throughout the study for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Naji Najib, B.Sc. Pharm, Study Director — IPRC Jordan; Abdullah Hiyari, MD, Principal Investigator — IPRC Jordan
Locations (1):
- International Pharmaceutical Research Center (IPRC), Amman, Jordan